CLINICAL TRIAL: NCT07366775
Title: Development of Telenursing for Diabetes Self-Management Education and Support (DSMES) Among Patients With Type 2 Diabetes Mellitus in Thailand: A Randomized Controlled Trial
Brief Title: A Telenursing Program to Support Diabetes Self-Management
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Ramida Subpaiboonkit, Principal Investigator, Lecturer, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2568-EXP092
Record Dates: First submitted 2026-01-07; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telenursing-Based DSMES Program (Experimental)
  Interventions: Behavioral: Telenursing-Based Diabetes Self-Management Education and Support
- Usual care (No Intervention): control group : receive usual care

INTERVENTIONS:
Behavioral: Telenursing-Based Diabetes Self-Management Education and Support — This intervention is a nurse-led, telenursing-based Diabetes Self-Management Education and Support (DSMES) program delivered over a 12-week period. It includes an initial face-to-face diabetes education session followed by scheduled follow-up sessions conducted via video calls. The program focuses on improving diabetes self-management through education, behavioral support, goal setting, problem-solving, and ongoing monitoring tailored to individual patient needs.
  Arms: Telenursing-Based DSMES Program

SUMMARY:
This randomized controlled trial aims to develop and evaluate a telenursing-based Diabetes Self-Management Education and Support (DSMES) program with uncontrolled type 2 diabetes mellitus in Thailand. The program is designed to improve diabetes self-management through nurse-led education, behavioral support, and regular follow-up delivered via telecommunication technologies.

Participants with type 2 diabetes and poor glycemic control will be randomly assigned to either an intervention group receiving a 12-week telenursing DSMES program or a control group receiving usual care. The intervention includes an initial in-person education session followed by structured video call follow-ups provided by nurse.

The primary outcome of this study is the feasibility of implementing telenursing for DSMES in Thailand. Secondary outcomes include changes in glycemic control, body mass index, diabetes knowledge, self-care behaviors, coping behaviors, quality of life, healthcare costs, and frequency of acute care use. The findings from this study are expected to provide evidence to support the use of telenursing as an accessible and sustainable approach for diabetes self-management in the Thai healthcare context.

ELIGIBILITY:
Inclusion Criteria:

* People with T2DM
* Adults (age 20-64) and older adults (65 and above)
* Uncontrolled diabetes, as determined by physician based on the diagnostic criteria of HbA1C > 7%
* Can read and write
* Own a smartphone
* Having internet connectivity
* Able to receive a video call or with assistance from a caregiver

Exclusion Criteria:

* Insulin-dependent patients
* Cognitive or mobility impairments , as assessed by the Thai Mental State Examination (TMSE). A TMSE score below 24 was considered indicative of cognitive impairment (The Nurse Association of Thailand, 2025).
* Requiring special nursing care, such as patients with severe diabetic complications or those who are bedridden.
* Previous extensive DSMES exposure

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2026-05-10 (Estimated); Study Completion 2026-05-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of telenursing for diabetes self-management education and support (DSMES) | at 12-week follow-up period after enrollment
  Feasibility outcomes, including participation rate, completion rate, and adherence level, were analyzed using descriptive statistics under the per-protocol (PP) approach, which included only participants who completed all study assessments.

SECONDARY OUTCOMES:
Glycated hemoglobin (HbA1c) level | From baseline to 12 weeks after enrollment
  HbA1c (%) will be measured using standard laboratory methods obtained from health assessment records. Change from baseline will be calculated as the difference between baseline and 12-week HbA1c values.
Body Mass Index (BMI) | From baseline to 12 weeks after enrollment
  Body mass index (kg/m²) will be calculated from measured weight and height obtained from health assessment records. Change from baseline will be calculated as the difference between baseline and 12-week BMI values.
Change from baseline in diabetes knowledge score measured by the Diabetes Knowledge Scale (DIAKS) | From baseline to 6 weeks and 12 weeks after enrollment
  Diabetes knowledge will be assessed using the Thai version of the Diabetes Knowledge Scale (DIAKS), consisting of 21 items with true, false, or don't know response options. Total scores will be calculated based on the number of correct responses. Change from baseline will be calculated using the 12-week assessment as the primary analysis time point; 6-week data will be used for interim descriptive analysis.
Self-care behavior | From baseline to 6 weeks and 12 weeks after enrollment
  Self-care behavior will be assessed using the Thai Diabetes Self-Management Questionnaire-Revised (T-DSMQ-R). Total scores will be calculated according to standard scoring procedures, with higher scores indicating better diabetes self-management. Change from baseline will be calculated using the 12-week assessment as the primary analysis time point; 6-week data will be used for interim descriptive analysis.
Positive coping behavior | From baseline to 6 weeks and 12 weeks after enrollment
  Positive coping behavior will be assessed using the Short Thai Stress Test (ST-5), a five-item questionnaire rated on a 0-3 Likert scale. Total scores range from 0 to 15, with higher scores indicating greater stress severity. Change from baseline will be calculated using the 12-week assessment as the primary analysis time point; 6-week data will be used for interim descriptive analysis.
Quality of life (QoL) | From baseline to 6 weeks and 12 weeks after enrollment
  Quality of life will be assessed using the Thai version of the Audit of Diabetes-Dependent Quality of Life (ADDQoL19). The average weighted impact (AWI) score will be calculated, with scores ranging from -9 to +3. Change from baseline will be calculated using the 12-week assessment as the primary analysis time point; 6-week data will be used for interim descriptive analysis.
Healthcare costs | at 12-week follow-up period after enrollment
  Healthcare costs will be assessed through review of medical and financial records, including outpatient visits, inpatient admissions, medications, laboratory tests, and other diabetes-related expenses. Total healthcare costs per participant will be summarized for the 12-week follow-up period.
Frequency of acute care use | at 12-week follow-up period after enrollment
  Frequency of acute care use will be assessed using hospital records, including emergency department visits and hospital admissions. The total number of acute care events per participant will be recorded during the follow-up period.
All-cause mortality | at 12-week follow-up period after enrollment
  All-cause mortality will be assessed using hospital follow-up records. Mortality status will be recorded for each participant during the follow-up period.